CLINICAL TRIAL: NCT03174106
Title: Longterm Follow-up of Cardiac Patients With an Smartphone-Application -A Randomized Clinical Study
Brief Title: Longterm Follow-up of Cardiac Patients With an Smartphone-Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Smartphone-application
Record Dates: First submitted 2017-05-19; First posted 2017-06-02 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Cardiac Rehabilitation; Mobile Health; Smartphone-application; Cardiac Disease; mHealth
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: Randomization to two different arms, intervention- or control-group
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The cardiologist, physical therapist and the physiologist at NIMI and Feiring will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone-Application (Experimental): Patients in "Smartphone-Application"-arm will get Access to the Application Vett, they will be learned how to use it. They will receive feedback based on their goals and tasks in the Application for one year, and they will also receive motivational Notifications through the Application, atleast once a week in the follow-up period. Patients in this arm will also have the possibility to send questions to their supervisor through the Application, in that case they will receive answer within two working days. In addition they will receive usual care which is described below.
  Interventions: Device: Smartphone-Application
- Control-group (No Intervention): Patients in the control-group will receive usual care consisting of general advice according to a heart-friendly lifestyle and follow-up by their general practitioner.

INTERVENTIONS:
Device: Smartphone-Application — Longterm follow-up after Cardiac rehabilitation With an Smartphone-Application
  Arms: Smartphone-Application

SUMMARY:
Cardiovascular disease is the leading cause of morbidity and mortality globally. Cardiac rehabilitation (CR) including exercise training are effective to reduce morbidity, mortality and risk factors such as physical fitness, cholesterol, triglycerides and blood pressure. The main goal for CR is to establish exercise training and other lifestyle changes as permanent changes in the patient's life. Many studies have shown that cardiac patients strive to maintain a heart-healthy lifestyle, one year after participating in CR. Furthermore, this leads to risk profile returning to the starting point where they got their Cardiac event. Changing a lifestyle is known to take time, and we believe that the patients need further follow-up beyond the time spent in traditional CR.

To our knowledge very few, if any, studies evaluates the use of modern technology in longterm follow-up focusing on maintaining a new lifestyle after participating in CR. The investigators would like to evaluate the effect of an dynamic application (app) with regard to physical fitness, lifestyle and quality of life (QoL), one year after CR. The investigators hypothesize that patients getting Access to a dynamic Application and tailored feedback through the application after CR will better be able to take care of physical Fitness and other lifestyle factors one year after CR, compared to patients getting usal care.

DETAILED DESCRIPTION:
Introduction:

Smartphones are widespread and in 2015 as much as 82% of the Norwegian population were owners of a smartphone. Recommendations has been pointed out in a new report from the Norwegian Board of Technology; health service should facilitate so that patients can follow up their health from home and simultaneously receive necessary help from the health service. The Norwegian Directorate of health points in a national action plan for e-health that evidence based digital tools in combination with an increase of competence will make it possible to reach health political goals such as quality levels, patient safety and an effective use of resources.

Across diseases adherence to treatment is one of the most important modifiable factors wich decreases the treatment effect. As much as 30-50% of patients do not adhere to recommended treatment. Adherence to treatment is complex and it depends on many factors; the patient, the patient surroundings (social support, the function of the health service, availability and resources) and characteristics with the disease and the corresponding treatment. World Health Organization (WHO) points to adherence to treatment as a global challenge and supports political decisions and research interventions that will increase adherence. Furthermore, adherence is considered to be a huge challenge in treatment for lifestyle changes such as smoking cessation, diet changes, training and physical activity. A meta-analysis (n=42 000) documented that "mixed mode of delivery interventions", where traditional techniques for behavior change was combined with digital tools, proved more effective than the use of traditional techniques for behavior change alone. Another meta-analysis (n=20 000) confirms this conclusion; therapy, guidance and conversation has an increased effect when it is used together with dedicated digital tools (6).

Cardiovascular disease is the leading cause of morbidity and mortality globally. Cardiac rehabilitation (CR) including exercise training are effective to reduce morbidity, mortality and modifiable risk factors such as physical fitness, cholesterol, triglycerides and blood pressure. The main goal for CR is to establish exercise training and other lifestyle changes as permanent changes in the patient's life. Many studies have shown that cardiac patients do not reach the therapeutic goals regarding secondary prophylaxis one year after participating in CR. In other words; patients are not able to maintain the new lifestyle after CR and their risk profile goes back to base. Changing a lifestyle is known to take time, and we believe that the patients need further follow-up beyond the time spent in traditional CR.

To our knowledge very few studies, if any, evaluates the use of modern technology aiming to help the patients to maintain a new lifestyle after participating in CR. The investigators would therefore like to implement a randomized clinical trial (RCT) to evaluate the effect of the dynamic Application Vett® With regard to physical Fitness (peak oxygen uptake), one year after CR.

Method:

* Design: The study will be a randomized clinical trial. Patients will be recruited from CR at Norwegian Institute of Sports Medicine (NIMI) and from Feiring. NIMI has an outpatient CR programme lasting for twelve weeks. Feiring has Institutional CR With two different durations at their programmes, whereas one of the programmes lasting four weeks an the other programme lasting for one week. The investigators will conduct a stratified randomization to ensure Equal number of patients from the different CR programmes into the intervention-group and the Control Group. Patients will be recruited when they finish CR.
* Intervention-group: In addition to usal care, patients in the intervention-group will get access to the application Vett®, as well as approximately one hour of training on how to use it and register personal goals together with study-coordinator. They will for a period of approximately twelve months have access to Vett® as well as personal follow-up through the app by a specialized physiotherapist. Vett® is an app developed by professor Kari Jorunn Kværner, doctor and specialist in cognitive training, guidance and counseling. Patients will be encouraged to set a minimum of two goals with associated tasks for the follow-up periode. Tasks will be the basis for reminders which the Application gives the patient. The patient decide when and how often reminders should come. The goals and tasks will be set according to the needs of each patient (individualized). The follow-up is individualized and dynamic and targets the patient under evaluation directly. Vett® makes it possible to create and set individual goals (e.g. exercise or eating fish) with tasks and reminders, weekly evaluation of the individual goals and ask questions to the supervisor. The application also gives the opportunity to receive tailored and motivational feedback from the supervisor. The supervisor has access to an administrator interface where it is possible to monitor what the patients are registering in relation to their personal goals and tasks, as well as sending tailored and motivational feedback. In this study, the patients will receive tailored feedback based on their achievements on personal goals and tasks through e-mail. They will receive feedback every week for the first Three months, then they will receive feedback as often as they want based on the conversation when included to the study. They will also receive 1-3 motivational feedbacks/notifications every week. Any questions to the supervisor will be answered by two working days. In the event of receiving health related questions (e.g changing of medication or chest pain) the patients will be advised to contact their general practitioner (GP). One year after CR patients will be called for a check-up, including questionnaires and a cardiorespiratory Fitness test.
* Control-Group: Patients in the control-group will receive what is current practice. In addition they will be called for a check-up, one year after entering CR, including questionnaires and a cardiorespiratory Fitness test. To day, usual care consist of advice regarding how to maintain their New lifestyle (exercise training, physical Activity and heart-healthy diet) and further follow-up by their GP.
* Power calculation: With a significant Level of 5%, Power of 0,80 and a effect size at 0,58 (Clinical important change as 3,5 ml/kg/min i VO2peak and a Standard deviation of 6 ml/kg/min), 48 patients is needed in each Group. With an estimated drop-out of 20%, 115 patients will be recruited to this study.
* Statistical analyzes: Both Parametric and non-Parametric analyzes will be used depending on the variables. Both intention-to-treat and per-protocol analyzes will be conducted in the effect-analyzes. T-test and variance analyzes will be used to investigate differences between Groups.

This study will provide New knowledge about the use of modern Technology with an Smartphone-Application in the follow-up of Cardiac patients. If the Application proves to be effective, this study will give clinicians a digital and evidence based tool for longterm follow-up of patients where changing lifestyle is the primary treatment.

ELIGIBILITY:
Inclusion Criteria:

* Finished Cardiac rehabilitation at NIMI or Feiring
* ≥ 40 years old
* Owner and user of a Smartphone
* Understanding basic Norwegian or English

Exclusion Criteria:

* Severe malignant disease that affects the patient's life to a greater extent than the heart disease
* Musculoskeletal- changes or diseases, that affect the patient's physical capacity and quality of life more than their heart disease
* Ischemia or arrytmia at treadmill test which gives the patient restrictions regarding exercise intensity equivalent >80% av HFmax eller BORG scale >15

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Change in Maximal oxygen consumption | Change from baseline to 12 months
  Physical capacity will be evaluated With maximal oxygen consumption. We will do a cardiorespiratory Fitness test on a treadmill With a standardized ramp-protocol and Direct measurement of oxygen consumption

SECONDARY OUTCOMES:
Change in Quality of Life | Change from baseline to 12 months
  Heart-Quality of Life (HeartQoL) will be used to assess quality of life. This is a disease specific questionnaire where you get an score between 0-3 (0 representing bad quality of life and 3 representing good quality of life). It consist of 14 question and you can get an emotional subscale and a physical subscale, aswell as a global scale.
Change in Quality of Life | Change from baseline to 12 months
  Euro Quality of life questionnaire (EQ-5D)
Change in Health Literacy | Change from baseline to 12 months
  European Health Literacy Survey questionnaire (HLS-EU-Q47)
Type D personality | Baseline
  Standard assessment of Negative Affectivity, Social Inhibition, and Type D personality (DS14).
Change in Endurance Fitness | Change from baseline to 12 months
  Time to exhaution, incline and speed at the treadmill test.

OTHER OUTCOMES:
Chang in Blood pressure | Change from baseline to 12 months
  Systolic and diastolic blood pressure, measured manually in resting sitting position before treadmill test
Change in Exercise habits | Change from baseline to 12 months
  The patients will be asked weekly exercise for the last year. Defined exercise as "at least 30 minutes of exercise With moderate to high intensity where you get sweaty and breathless"

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - LHL-Feiring, Feiring
  - NIMI, Oslo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lunde P, Bye A, Grimsmo J, Pripp AH, Ritschel V, Jarstad E, Nilsson BB. Effects of Individualized Follow-Up With an App Postcardiac Rehabilitation: Five-Year Follow-Up of a Randomized Controlled Trial. J Med Internet Res. 2025 Feb 13;27:e60256. doi: 10.2196/60256. PMID 39946716
- [Derived] Lunde P, Bye A, Bergland A, Nilsson BB. Effects of individualized follow-up with a smartphone-application after cardiac rehabilitation: protocol of a randomized controlled trial. BMC Sports Sci Med Rehabil. 2019 Nov 21;11:34. doi: 10.1186/s13102-019-0148-2. eCollection 2019. PMID 31768261